CLINICAL TRIAL: NCT01849627
Title: Eat Well for Life: A Weight Loss Maintenance Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9141B
Record Dates: First submitted 2013-04-30; First posted 2013-05-08 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: weight loss maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-ED (Experimental): This condition will focus lowering on the energy density of the diet of the diet. This prescription does not include goals for any other nutrients, thus there are no energy goals.
  Interventions: Behavioral: Low-ED
- Energy Balance (Experimental): This condition will focus have an energy balance prescription. Participants will be asked to consume a daily energy intake at estimated energy needs for weight loss maintenance.
  Interventions: Behavioral: Energy Balance

INTERVENTIONS:
Behavioral: Low-ED — This condition will be instructed to make food consumption decisions based solely upon the ED of a food. The goal of the ED condition will be to consume at least 10 foods ≤ 1.0 kcal/g (i.e., fruits and vegetables, broth based soups, non-fat yogurts, some legumes, egg substitutes, some white fish, etc.) and no more than 2 foods ≥ 3.0 kcal/g (i.e., crackers, chips, cookies, hard cheeses, hot dogs, salad dressings, etc.) per day.
  Arms: Low-ED
Behavioral: Energy Balance — Energy Balance will receive an individualized daily energy goal which will be their measured resting metabolic rate multiplied by a physical activity level (PAL) of 1.12 (men) or 1.14 (women) (low active).
  Arms: Energy Balance

SUMMARY:
A study to investigate the effect of a low-ED prescription (consume ≥10 foods ≤ 1.0 kcal/g and ≤ 2 foods ≥ 3.0 kcal/g per day) versus an energy balance prescription (consume a daily energy intake at estimated energy needs for maintenance) on weight loss maintenance.

DETAILED DESCRIPTION:
Obesity increases the risk of several health conditions. Weight loss of 5-10% of initial weight reduces the risk of several diseases. This degree of weight loss is achievable in behavioral obesity programs. However, about 33% of initial weight loss is regained within one year and very little weight loss is maintained within three to five years. Thus, new strategies improving long-term weight loss maintenance are needed. One dietary strategy that increases self-reported satiation and satiety is consuming a low energy density (ED) diet. A low-ED diet allows a greater weight of food relative to total energy to be consumed, which is the proposed mechanism for the enhanced self-reported satiation and satiety found with low-ED meals. Research has shown that when participants are served low-ED meals, while total weight of food consumed does not change, meal energy intake decreases. Importantly, when low-ED meals are consumed across several days, reduced energy intake continues to occur, showing no degree of energy intake compensation. To address the gaps regarding the relationship between dietary ED and weight loss maintenance, we propose to conduct a randomized controlled trial (RCT) examining the effect of a low-ED prescription and its proposed mechanisms on weight loss maintenance.

The primary hypotheses are:

1. Low-ED will have less weight regain than Energy Balance at 22 months.

   a. Weight regain at 10, 16, and 22 months will be examined to determine if differences occur between conditions.
2. Low-ED will consume a lower ED diet, less energy and percent energy from fat, and greater grams from solid food and fiber than Energy Balance at 10, 16, and 22 months.

   The secondary hypotheses are:
3. Identify mechanisms (mediators) by which reducing ED improves long-term lower energy intake, thus:

   1. Low-ED will self-report lower hunger and greater satiation and satiety during EMA than Energy Balance at 10, 16, and 22 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Body mass index (BMI) between 27 and 45 kg/m2

Exclusion Criteria:

* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Individuals reporting joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate
* Report being unable to walk for 2 blocks (1/4 mile) without stopping
* Report major psychiatric diseases or organic brain syndromes.
* Are currently participating in a weight loss program and/or taking weight loss or appetite regulation medication or lost > 5% of body weight during the past 6 months
* Have had bariatric surgery for weight loss or are planning to have bariatric surgery in the next 22 months
* Intend to move outside of the metropolitan area within the time frame of the investigation
* Are pregnant, lactating, < 6 months post-partum, or plan to become pregnant during the investigation
* Report not being able to consume meal replacements

To participate in the weight loss maintenance phase, participants will need to lose equal to or greater than 8% of their body weight from the baseline measure at the conclusion of the 4-month weight loss phase.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Anthropometrics from Baseline at 4, 10, 16, and 22 months | 0, 4, 10, 16, and 22 months
  Height, weight, and BMI will be assessed.
Changes in diet from baseline at 4, 10, 16, and 22 months | 0, 4, 10, 16, and 22 months
  Three day food records will be used to assess energy, grams, energy density, macronutrients, fiber, and food group servings.

SECONDARY OUTCOMES:
Changes in hunger, satiation, and satiety from baseline at 4, 10, 16, and 22 months | 0, 4, 10, 16, and 22 months
  Changes in EMA measures on hunger, satiation, and satiety will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, LDN, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Engelgau MM, Geiss LS, Saaddine JB, Boyle JP, Benjamin SM, Gregg EW, Tierney EF, Rios-Burrows N, Mokdad AH, Ford ES, Imperatore G, Narayan KM. The evolving diabetes burden in the United States. Ann Intern Med. 2004 Jun 1;140(11):945-50. doi: 10.7326/0003-4819-140-11-200406010-00035. PMID 15172919
- [Background] Field AE, Coakley EH, Must A, Spadano JL, Laird N, Dietz WH, Rimm E, Colditz GA. Impact of overweight on the risk of developing common chronic diseases during a 10-year period. Arch Intern Med. 2001 Jul 9;161(13):1581-6. doi: 10.1001/archinte.161.13.1581. PMID 11434789
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] Neter JE, Stam BE, Kok FJ, Grobbee DE, Geleijnse JM. Influence of weight reduction on blood pressure: a meta-analysis of randomized controlled trials. Hypertension. 2003 Nov;42(5):878-84. doi: 10.1161/01.HYP.0000094221.86888.AE. Epub 2003 Sep 15. PMID 12975389
- [Background] Klein S, Burke LE, Bray GA, Blair S, Allison DB, Pi-Sunyer X, Hong Y, Eckel RH; American Heart Association Council on Nutrition, Physical Activity, and Metabolism. Clinical implications of obesity with specific focus on cardiovascular disease: a statement for professionals from the American Heart Association Council on Nutrition, Physical Activity, and Metabolism: endorsed by the American College of Cardiology Foundation. Circulation. 2004 Nov 2;110(18):2952-67. doi: 10.1161/01.CIR.0000145546.97738.1E. Epub 2004 Oct 27. PMID 15509809
- [Background] Pi-Sunyer FX. How effective are lifestyle changes in the prevention of type 2 diabetes mellitus? Nutr Rev. 2007 Mar;65(3):101-10. doi: 10.1111/j.1753-4887.2007.tb00287.x. PMID 17425061
- [Background] Foster GD, Makris AP, Bailer BA. Behavioral treatment of obesity. Am J Clin Nutr. 2005 Jul;82(1 Suppl):230S-235S. doi: 10.1093/ajcn/82.1.230S. PMID 16002827
- [Background] Wadden TA, Crerand CE, Brock J. Behavioral treatment of obesity. Psychiatr Clin North Am. 2005 Mar;28(1):151-70, ix. doi: 10.1016/j.psc.2004.09.008. No abstract available. PMID 15733617
- [Background] Jeffery RW, Drewnowski A, Epstein LH, Stunkard AJ, Wilson GT, Wing RR, Hill DR. Long-term maintenance of weight loss: current status. Health Psychol. 2000 Jan;19(1S):5-16. doi: 10.1037/0278-6133.19.suppl1.5. PMID 10709944
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Havel PJ. Peripheral signals conveying metabolic information to the brain: short-term and long-term regulation of food intake and energy homeostasis. Exp Biol Med (Maywood). 2001 Dec;226(11):963-77. doi: 10.1177/153537020122601102. PMID 11743131
- [Background] Karhunen L, Lyly M, Lapvetelainen A, Kolehmainen M, Laaksonen DE, Lahteenmaki L, Poutanen K. Psychobehavioural factors are more strongly associated with successful weight management than predetermined satiety effect or other characteristics of diet. J Obes. 2012;2012:274068. doi: 10.1155/2012/274068. Epub 2012 Jun 25. PMID 22792447
- [Background] Ebbeling CB, Swain JF, Feldman HA, Wong WW, Hachey DL, Garcia-Lago E, Ludwig DS. Effects of dietary composition on energy expenditure during weight-loss maintenance. JAMA. 2012 Jun 27;307(24):2627-34. doi: 10.1001/jama.2012.6607. PMID 22735432
- [Background] Rolls BJ, Drewnowski A, Ledikwe JH. Changing the energy density of the diet as a strategy for weight management. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S98-103. doi: 10.1016/j.jada.2005.02.033. PMID 15867904
- [Background] Rolls BJ. The relationship between dietary energy density and energy intake. Physiol Behav. 2009 Jul 14;97(5):609-15. doi: 10.1016/j.physbeh.2009.03.011. Epub 2009 Mar 20. PMID 19303887
- [Background] Perez-Escamilla R, Obbagy JE, Altman JM, Essery EV, McGrane MM, Wong YP, Spahn JM, Williams CL. Dietary energy density and body weight in adults and children: a systematic review. J Acad Nutr Diet. 2012 May;112(5):671-84. doi: 10.1016/j.jand.2012.01.020. Epub 2012 Apr 3. PMID 22480489
- [Background] Rolls BJ. Plenary Lecture 1: Dietary strategies for the prevention and treatment of obesity. Proc Nutr Soc. 2010 Feb;69(1):70-9. doi: 10.1017/S0029665109991674. Epub 2009 Dec 3. PMID 19954563
- [Background] Rolls BJ, Roe LS, Meengs JS. Reductions in portion size and energy density of foods are additive and lead to sustained decreases in energy intake. Am J Clin Nutr. 2006 Jan;83(1):11-7. doi: 10.1093/ajcn/83.1.11. PMID 16400043
- [Background] Ello-Martin JA, Ledikwe JH, Rolls BJ. The influence of food portion size and energy density on energy intake: implications for weight management. Am J Clin Nutr. 2005 Jul;82(1 Suppl):236S-241S. doi: 10.1093/ajcn/82.1.236S. PMID 16002828
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Lowe MR, Tappe KA, Annunziato RA, Riddell LJ, Coletta MC, Crerand CE, Didie ER, Ochner CN, McKinney S. The effect of training in reduced energy density eating and food self-monitoring accuracy on weight loss maintenance. Obesity (Silver Spring). 2008 Sep;16(9):2016-23. doi: 10.1038/oby.2008.270. PMID 18483475
- [Background] Raynor HA, Van Walleghen EL, Bachman JL, Looney SM, Phelan S, Wing RR. Dietary energy density and successful weight loss maintenance. Eat Behav. 2011 Apr;12(2):119-25. doi: 10.1016/j.eatbeh.2011.01.008. Epub 2011 Jan 25. PMID 21385641
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Bachman JL, Raynor HA. Effects of manipulating eating frequency during a behavioral weight loss intervention: a pilot randomized controlled trial. Obesity (Silver Spring). 2012 May;20(5):985-92. doi: 10.1038/oby.2011.360. Epub 2011 Dec 15. PMID 22173575
- [Background] Raynor HA, Looney SM, Steeves EA, Spence M, Gorin AA. The effects of an energy density prescription on diet quality and weight loss: a pilot randomized controlled trial. J Acad Nutr Diet. 2012 Sep;112(9):1397-1402. doi: 10.1016/j.jand.2012.02.020. Epub 2012 May 9. PMID 22575072
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Thomas S, Reading J, Shephard RJ. Revision of the Physical Activity Readiness Questionnaire (PAR-Q). Can J Sport Sci. 1992 Dec;17(4):338-45. PMID 1330274
- [Background] Ribisl PM, Lang W, Jaramillo SA, Jakicic JM, Stewart KJ, Bahnson J, Bright R, Curtis JF, Crow RS, Soberman JE; Look AHEAD Research Group. Exercise capacity and cardiovascular/metabolic characteristics of overweight and obese individuals with type 2 diabetes: the Look AHEAD clinical trial. Diabetes Care. 2007 Oct;30(10):2679-84. doi: 10.2337/dc06-2487. Epub 2007 Jul 20. PMID 17644623
- [Background] Look AHEAD Research Group; Wadden TA, West DS, Delahanty L, Jakicic J, Rejeski J, Williamson D, Berkowitz RI, Kelley DE, Tomchee C, Hill JO, Kumanyika S. The Look AHEAD study: a description of the lifestyle intervention and the evidence supporting it. Obesity (Silver Spring). 2006 May;14(5):737-52. doi: 10.1038/oby.2006.84. PMID 16855180
- [Background] Ryan DH, Espeland MA, Foster GD, Haffner SM, Hubbard VS, Johnson KC, Kahn SE, Knowler WC, Yanovski SZ; Look AHEAD Research Group. Look AHEAD (Action for Health in Diabetes): design and methods for a clinical trial of weight loss for the prevention of cardiovascular disease in type 2 diabetes. Control Clin Trials. 2003 Oct;24(5):610-28. doi: 10.1016/s0197-2456(03)00064-3. PMID 14500058
- [Background] Wing RR, Tate DF, Gorin AA, Raynor HA, Fava JL. A self-regulation program for maintenance of weight loss. N Engl J Med. 2006 Oct 12;355(15):1563-71. doi: 10.1056/NEJMoa061883. PMID 17035649
- [Background] Wing RR. Behavioral approaches to the treatment of obesity. In: Bray GA, Bouchard C, James WPT, eds. Handbook of Obesity. New York: Marcel Dekker, Inc.; 1998:855-873
- [Background] Jakicic JM, Clark K, Coleman E, Donnelly JE, Foreyt J, Melanson E, Volek J, Volpe SL; American College of Sports Medicine. American College of Sports Medicine position stand. Appropriate intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2001 Dec;33(12):2145-56. doi: 10.1097/00005768-200112000-00026. PMID 11740312
- [Background] Malik VS, Schulze MB, Hu FB. Intake of sugar-sweetened beverages and weight gain: a systematic review. Am J Clin Nutr. 2006 Aug;84(2):274-88. doi: 10.1093/ajcn/84.1.274. PMID 16895873
- [Background] Flood-Obbagy JE, Rolls BJ. The effect of fruit in different forms on energy intake and satiety at a meal. Appetite. 2009 Apr;52(2):416-22. doi: 10.1016/j.appet.2008.12.001. Epub 2008 Dec 6. PMID 19110020
- [Background] Rolls BJ. The Volumetrics Eating Plan. New York: HarperCollins Publisher; 2005.
- [Background] Ard JD, Fitzpatrick S, Desmond RA, Sutton BS, Pisu M, Allison DB, Franklin F, Baskin ML. The impact of cost on the availability of fruits and vegetables in the homes of schoolchildren in Birmingham, Alabama. Am J Public Health. 2007 Feb;97(2):367-72. doi: 10.2105/AJPH.2005.080655. Epub 2006 Nov 30. PMID 17138914
- [Background] Hipskind P, Glass C, Charlton D, Nowak D, Dasarathy S. Do handheld calorimeters have a role in assessment of nutrition needs in hospitalized patients? A systematic review of literature. Nutr Clin Pract. 2011 Aug;26(4):426-33. doi: 10.1177/0884533611411272. PMID 21775638
- [Background] McDoniel SO. Systematic review on use of a handheld indirect calorimeter to assess energy needs in adults and children. Int J Sport Nutr Exerc Metab. 2007 Oct;17(5):491-500. doi: 10.1123/ijsnem.17.5.491. PMID 18046058
- [Background] Gerrior S, Juan W, Basiotis P. An easy approach to calculating estimated energy requirements. Prev Chronic Dis. 2006 Oct;3(4):A129. Epub 2006 Sep 15. PMID 16978504
- [Background] Brantley P, Appel L, Hollis J, Stevens V, Ard J, Champagne C, Elmer P, Harsha D, Myers V, Proschan M, William V, Svetkey L. Design considerations and rationale of a multi-center trial to sustain weight loss: the Weight Loss Maintenance Trial. Clin Trials. 2008;5(5):546-56. doi: 10.1177/1740774508096315. PMID 18827047
- [Background] Delbridge EA, Prendergast LA, Pritchard JE, Proietto J. One-year weight maintenance after significant weight loss in healthy overweight and obese subjects: does diet composition matter? Am J Clin Nutr. 2009 Nov;90(5):1203-14. doi: 10.3945/ajcn.2008.27209. Epub 2009 Sep 30. PMID 19793858
- [Background] Borushek A. The CalorieKing. Cost Mesa: Family Health Publications; 2010.
- [Background] Lohman TR, Roche AF, Martorell R. Anthropometric Standardization Reference Manual. Champaign,Illinois: Human Kinetics Books; 1988.
- [Background] Paffenbarger RS Jr, Hyde RT, Wing AL, Lee IM, Jung DL, Kampert JB. The association of changes in physical-activity level and other lifestyle characteristics with mortality among men. N Engl J Med. 1993 Feb 25;328(8):538-45. doi: 10.1056/NEJM199302253280804. PMID 8426621
- [Background] Rauh MJ, Hovell MF, Hofstetter CR, Sallis JF, Gleghorn A. Reliability and validity of self-reported physical activity in Latinos. Int J Epidemiol. 1992 Oct;21(5):966-71. doi: 10.1093/ije/21.5.966. PMID 1468861
- [Background] Munsch S, Meyer AH, Milenkovic N, Schlup B, Margraf J, Wilhelm FH. Ecological momentary assessment to evaluate cognitive-behavioral treatment for binge eating disorder. Int J Eat Disord. 2009 Nov;42(7):648-57. doi: 10.1002/eat.20657. PMID 19197978
- [Background] Barnard ND, Scialli AR, Bertron P, Hurlock D, Edmonds K. Acceptability of a therapeutic low-fat, vegan diet in premenopausal women. Journal of Nutrition Education 2000;32:314-319.
- [Background] Ebbeling CB, Leidig MM, Feldman HA, Lovesky MM, Ludwig DS. Effects of a low-glycemic load vs low-fat diet in obese young adults: a randomized trial. JAMA. 2007 May 16;297(19):2092-102. doi: 10.1001/jama.297.19.2092. PMID 17507345
- [Background] Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: Wiley & Sons; 1987.
- [Background] Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Arch Gen Psychiatry. 2002 Oct;59(10):877-83. doi: 10.1001/archpsyc.59.10.877. PMID 12365874
- [Background] Holmbeck GN. Post-hoc probing of significant moderational and mediational effects in studies of pediatric populations. J Pediatr Psychol. 2002 Jan-Feb;27(1):87-96. doi: 10.1093/jpepsy/27.1.87. PMID 11726683
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406